CLINICAL TRIAL: NCT02938975
Title: Field Efficacy Of Insecticide Treated Uniforms And Skin Repellents To Reduce Malaria Incidence In Military Personnel On Active Duty In Regions Of Hyperendemicity
Brief Title: Field Efficacy Of Insecticide Treated Uniforms And Skin Repellents for Malaria Prevention
Acronym: URCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ifakara Health Institute (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BIT014 PR001 V01
Record Dates: First submitted 2016-08-05; First posted 2016-10-19 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Malaria
Keywords: malaria; personal protection; permethrin treated clothing; insect repellents; army personnel; cluster randomised trial
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): placebo group receiving untreated army combat uniform and placebo lotion. Assigned interventions: Placebo lotion - a liposome lotion with no DEET Army combat uniform - army combat uniform with no permethrin
  Interventions: Other: Placebo lotion; Other: Army combat uniform
- Combo (Active Comparator): Combined intervention group of receiving Permethrin treated uniform 0.52% w/w and 30% DEET liposome formula.
  Ultra 30 Insect Repellent Lotion (30% Lipo DEET) One application of Lipo DEET protects for up to 12 hours. DEET is a broad spectrum insect repellent that has been extensively tested for safety and toxicity for human use and its efficacy against a broad variety of arthropod vectors.
  Permethrin Factory-Treated Army Combat Uniforms treated by the military apparel contractor Warmkraft Permethrin is considered the most effective clothing treatment available to prevent insect bites through fabric. The Army objective is to provide 90% bite protection for at least 50 launderings.
  Interventions: Other: Ultra 30 Insect Repellent Lotion (30% Lipo DEET); Other: Permethrin Factory-Treated Army Combat Uniforms
- Permethrin (Active Comparator): permethrin intervention group receiving Permethrin treated uniform 0.52% w/w and placebo lotion.
  Permethrin Factory-Treated Army Combat Uniforms treated by the military apparel contractor Warmkraft
  Placebo lotion: liposome lotion with no DEET
  Interventions: Other: Permethrin Factory-Treated Army Combat Uniforms; Other: Placebo lotion
- DEET (Active Comparator): DEET intervention group receiving untreated army combat uniform and 30% DEET liposome formula.
  Ultra 30 Insect Repellent Lotion (30% Lipo DEET) Army combat uniform with no permethrin
  Interventions: Other: Ultra 30 Insect Repellent Lotion (30% Lipo DEET); Other: Army combat uniform

INTERVENTIONS:
Other: Ultra 30 Insect Repellent Lotion (30% Lipo DEET) — One application of Lipo DEET protects for up to 12 hours and has a pleasant odour and non-greasy "feel" on the skin. DEET is a broad spectrum insect repellent and was selected this study because it has been extensively tested for safety and toxicity for human use and its efficacy against a broad variety of arthropod vectors. DEET was first registered in 1957 and has been conclusively proven to be safe for use on adults, children, pregnant and lactating mothers.
  This Liposome-based repellent is the newest advancement in insect repellent technology. The Liposome envelops the active ingredient, DEET, and slowly time-releases it as needed, thereby extending the effectiveness of the repellent and reducing dermal absorption.
  Arms: Combo; DEET
Other: Permethrin Factory-Treated Army Combat Uniforms — Permethrin is the U.S., Australian and United Kingdom (UK) military's standard repellent for application to fabric and is considered the most effective clothing treatment available to prevent insect bites through fabric. The Army objective is to provide 90% bite protection for at least 50 launderings; an objective easily met through factory treatment of uniforms, which demonstrates 99-100% bite protection up to 50 launderings (the expected lifetime of the uniform).
  Arms: Combo; Permethrin
Other: Placebo lotion — A liposome lotion with no DEET
  Arms: Permethrin; Placebo
Other: Army combat uniform — Army combat uniform with no permethrin
  Arms: DEET; Placebo

SUMMARY:
Purpose

While there is strong evidence that permethrin treated clothing prevents insect bites there is insufficient evidence from trials to demonstrate a reduction in infections. The evidence that topical insect repellants prevent malaria is more robust, but studies in civilian suffer from poor compliance. It is not known if there is an added benefit from combining the two. The effectiveness of permethrin-treated uniforms with and without DEET lotion are compared in a 2x2 design in Mgambo Jeshi la Kujenga Taifa (JKT) military camp in Tanga region.

The four arms are: 1) combined intervention group receiving permethrin treated uniform (PTU) and 30% DEET (diethyl toluamide) liposome formula; 2) permethrin intervention group receiving PTU and placebo lotion; 3) DEET intervention group receiving untreated army combat uniform (ACU) and 30% DEET liposome formula; 4) placebo group receiving untreated ACU and placebo lotion. Both participants and investigators will be blinded to treatment allocation.

The outcome measure is the incidence of Plasmodium falciparum malaria infection measured by Polymerase Chain Reaction every month by active case detection.

DETAILED DESCRIPTION:
The study is a prospective, cluster-randomised placebo controlled trial using a 4-arm non-inferiority design with 12 months of follow-up. Healthy recruits of the Tanzanian National Service Program JKT Mgambo Camp will be enrolled in the trial. The recruits come from all over Tanzania. The transmission in the camp is relatively high: the incidence of malaria infection in Mgambo camp among recruits in the last quarter of 2014 was 0.68 per person per year measured by RDT.

One thousand five hundred recruits will be enrolled in the trial. Randomisation will be based on combania (the company, comprising typically 30-50 recruits). Recruits in a combania perform all activities together as a group. The randomisation will be unequal since the investigators expect that the primary comparison requiring the greatest precision is that of adding DEET lotion to PTU. Investigators will randomise 500 recruits for each arm of the primary comparison (PTU plus DEET, PTU uniform only) and 250 recruits to each of DEET only and placebo.

Compliance will be maximised by requesting participants to use their uniforms and lotions only at night. Monitoring of uniform use will be conducted by random spot checks of participants in the evenings by study staff. In addition, bottles of lotion will be weighed on a monthly basis during active case detection as a direct measure of compliance with lotion use.

Artemether-lumefantrine (Co-Artem) will be given to any participant with a temperature of ≥37.5 degrees centigrade or a history of fever in the past 48h, and P. falciparum parasites detected by RDT in the absence of other detectable cause of fever.

The participants' activities for the previous two weeks will be recorded by questionnaire by study staff during active case detection. Time away from the camp or in the sick bay and prophylactic periods in the case of antimalarial treatment will be excluded from time at risk.

Soldiers are a vulnerable group because they have limited ability to protect their own interests. It is therefore, particularly important that they should be prevented from being involved in the research project because they feel it is their duty to do so or that they may be subject to penalty from senior members of the army. Therefore, in order to protect the soldiers from coercion the ethical review process for the research is conducted the same processes procedure as is required by a civilian Institutional Review Board (IRB). In addition, service members' commanders or supervisors may not be in the room during the consent process. It will be stressed to Tanzania People's Defence Force (TPDF) staff performing spot checks that they are merely to monitor compliance and should not coerce participants into wearing their uniforms when in the barracks

ELIGIBILITY:
Inclusion Criteria:

Member of a platoon passes physical examination - no underlying health risks females that are not pregnant malaria negative at enrolment consents to participate

Exclusion Criteria:

Not assigned to a platoon underlying health risks - does not pass physical examination pregnant female (pregnant females are not recruited into the army) malaria positive at enrolment does not consent to participate

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1500 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Plasmodium falciparum malaria through monthly measurement of malaria positivity by direct polymerase chain reaction (PCR) to detect parasite DNA | Monthly active case detection for 12 months
  Blood spots will be collected on Whatman 3 filter paper and processed for PCR detection of parasites

SECONDARY OUTCOMES:
Incidence of clinical malaria through monthly measurement malaria positivity of SD Bioline Malaria Rapid Diagnostic Test to test for parasite antigen | Active and passive case detection for 12 months
  Both active and passive malaria case detection will be taken by malaria RDT (SD Bioline Malaria Incidence of RDT positivity Participants will be tested for malaria every month using Rapid Diagnostic Test (RDT) SD Bioline Malaria Antigen Pf/Pan (SD RDT) with RDT results interpreted by the Deki Reader device.
Compliance with intervention as measured through spot checking and weighing of repellent bottles | Monthly assessment of intervention compliance with uniforms and lotions provided for 12 months
  Each month bottles of repellent or placebo lotion will be weighed to measure application of repellent. Compliance with uniforms will be observed by spot checks once a month.
Protective efficacy of uniforms measured by reduction in Anopheles arabiensis bites among those wearing uniforms for a sub-sample of uniforms tested under laboratory conditions with free flying mosquitoes | After 12 months
  A random sample of 100 uniforms will be tested in the laboratory at the end of the study to measure their efficacy in preventing mosquito bites.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Moore, PhD, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute, Bagamoyo, Tanzania

REFERENCES:
- [Derived] Msellemu D, Ross A, Temu L, Moshi I, Hofer L, Mwanziva C, Kohi YM, Moore SJ. Effect of interventions to reduce malaria incidence among military personnel on active duty: study protocol for a cluster randomised controlled trial of the impact of etofenprox-treated uniforms, permethrin-treated uniforms and DEET insect repellent. Trials. 2021 Nov 21;22(1):825. doi: 10.1186/s13063-021-05801-9. PMID 34802455